CLINICAL TRIAL: NCT01539226
Title: A Multi-Centre, Randomised, Double-Blind, Placebo-Controlled Safety and Efficacy Trial of a Dapivirine Vaginal Matrix Ring in Healthy HIV-Negative Women
Brief Title: Safety and Efficacy Trial of a Dapivirine Vaginal Matrix Ring in Healthy HIV-Negative Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM 027
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Results first posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-07

CONDITIONS: HIV Infections
Keywords: HIV Infections; Anti-HIV agents; HIV-1
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Vaginal Ring (Placebo Comparator): Vaginal Ring containing 0.0 mg Dapivirine
  Interventions: Combination Product: Placebo Vaginal Ring
- Dapivirine Vaginal Ring (Experimental): Vaginal Ring containing 25mg of Dapivirine
  Interventions: Combination Product: Dapivirine Vaginal Ring, 25 mg

INTERVENTIONS:
Combination Product: Placebo Vaginal Ring — Dapivirine Vaginal Ring containing 0.0 mg of dapivirine
  Arms: Placebo Vaginal Ring
Combination Product: Dapivirine Vaginal Ring, 25 mg — Dapivirine Vaginal Ring containing 25 mg of dapivirine
  Arms: Dapivirine Vaginal Ring

SUMMARY:
This is a double-blind, randomised, placebo-controlled study to assess the safety and efficacy of a silicone elastomer vaginal matrix ring.

DETAILED DESCRIPTION:
A multi center, randomized, double-blind, placebo=controlled safety and efficacy trial of a Dapivirine Vaginal Matrix Ring in healthy HIV-negative women.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 and < 45 years of age, at screening, who can provide informed consent;
* Available for all visits and consent to follow all procedures scheduled for the trial;
* Self-reported sexually active (defined as an average of at least one penetrative penile-vaginal coital act per month for the last 3 months prior to screening);
* HIV-negative as determined by the HIV algorithm applied at screening and enrolment;
* On a stable form of contraception as defined within section 5.4 and willing to continue on stable contraception for the duration of the clinical trial, unless post-menopausal or surgically sterilised;
* Asymptomatic for genital infections at the time of enrolment (if a woman is diagnosed with any clinically significant curable STI, she must have initiated treatment at least 1 week prior to enrolment and have completed the full course of treatment);
* Willing to provide adequate locator information for trial retention purposes and be reachable per local standard procedures (e.g., by home visit or telephone; or via family or close neighbour contacts); confidentiality to be maintained;
* Willing to refrain from participation in another research trial using drugs, vaccines, medical devices, microbicides or oral pre-exposure prophylaxis investigational drugs for the duration of the IPM 027 trial.

Exclusion Criteria:

* Currently pregnant or last pregnancy within 3 months prior to screening or intends to become pregnant during trial participation;
* Currently breast-feeding;
* Non-therapeutic injection drug use in the 12 months prior to screening;
* Participated in another research trial using drugs, medical devices, microbicides or oral pre-exposure prophylaxis agents within 60 days prior to screening;
* Previously participated or currently participating in any HIV vaccine trial;
* Untreated, clinically significant urogenital infections , e.g., urinary tract, or other sexually transmitted infections, or other gynaecological symptoms within 1 week prior to enrolment;
* Has a Grade 2 or higher pelvic examination finding, according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events; Addendum 1 Female Genital Grading Table for Use in Microbicide Studies;
* History of significant urogenital or uterine prolapse, undiagnosed vaginal bleeding, diagnosed chronic and/or recurrent vulvovaginal candidiasis, urethral obstruction, incontinence or urge incontinence;
* Any gynaecological surgery within 90 days prior to screening;
* Any Grade 1 or higher baseline aspartate aminotransferase (AST), alanine transaminase (ALT), or platelet count, and any Grade 2 or higher baseline haematology, chemistry or urinalysis laboratory value according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events;
* Any history of anaphylaxis or severe allergy resulting in angioedema; or a history of sensitivity/allergy to latex or a silicone elastomer;
* Any history of diabetes mellitus and chronic use of oral corticosteroid therapy; and any uncontrolled serious chronic or progressive disease;
* Cervical cytology at screening that requires cryotherapy, biopsy or treatment (other than for infection). Women with Grade 1 cervical cytology findings can be enrolled upon completion of the initial phase of evaluation if no current treatment is indicated (based on local standard of care for management of abnormal cervical cytology);
* Any condition(s) that, in the opinion of the investigator, might put the participant at risk, or interfere with the trial objectives or the participant's adherence to trial requirements.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1959 (Actual)
Dates: Start 2012-03-27 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annalene Nel, Study Director — Beijing Immupeutics Medicine Technology Limited
Locations (7):
- South Africa (6):
  - Qhakaza Mbokodo, Ladysmith, KwaZulu-Natal
  - Prevention of HIV / AIDS (PHIVA) Project, Pinetown, KwaZulu-Natal
  - Ndlovu Medical Centre, Elandsdoorn, Limpopo
  - Madibeng Centre for Research (MCR), Brits
  - Desmond Tutu HIV Foundation, Guinea Fowl Road, Sunnydale, Fish Hoek, Cape Town
  - Maternal, Adolescent and Child Health (MatCH), Plessislaer
- MRC/UVRI Uganda Research Unit on AIDS, Plot 51-59, Nakiwogo Road, PO BOX 49, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kusemererwa S, Ruzagira E, Onyango M, Kabarambi A, Abaasa A. Associations between intravaginal practices and incidence of sexually transmitted infections and bacterial vaginosis among women enrolled in the dapivirine vaginal ring trial (The Ring Study) in southwestern Uganda: a retrospective secondary analysis. BMJ Open. 2024 Apr 8;14(4):e079497. doi: 10.1136/bmjopen-2023-079497. PMID 38589266
- [Derived] Steytler J, Craig C, van der Ryst E, Van Baelen B, Nuttall J, van Niekerk N, Mellors J, Parikh U, Wallis C; Ring Study and the DREAM Trial Study Teams. Characterization of Viruses in Phase 3 and Phase 3b Trials (the Ring Study and the Dapivirine Ring Extended Access and Monitoring Trial) of the Dapivirine Vaginal Ring for Human Immunodeficiency Virus Type 1 Infection Risk Reduction. Clin Infect Dis. 2023 Mar 21;76(6):996-1002. doi: 10.1093/cid/ciac875. PMID 36345569
- [Derived] Kusemererwa S, Abaasa A, Kabarambi A, Onyango M, Mugisha JO. Assessment of risk compensation following use of the dapivirine vaginal ring in southwestern Uganda. Sex Transm Infect. 2022 Feb;98(1):32-37. doi: 10.1136/sextrans-2020-054718. Epub 2021 Feb 4. PMID 33542153
- [Derived] Kusemererwa S, Abaasa A, Onyango M, Nel AM, Isaacs M, Asiki G. Contraceptive Preference Among Women at Risk of HIV Acquisition in a Preparatory Screening Study for a Phase III Microbicide Trial in South Western Uganda. AIDS Behav. 2018 Jul;22(Suppl 1):131-138. doi: 10.1007/s10461-018-2177-3. PMID 29855975
- [Derived] Nel A, van Niekerk N, Kapiga S, Bekker LG, Gama C, Gill K, Kamali A, Kotze P, Louw C, Mabude Z, Miti N, Kusemererwa S, Tempelman H, Carstens H, Devlin B, Isaacs M, Malherbe M, Mans W, Nuttall J, Russell M, Ntshele S, Smit M, Solai L, Spence P, Steytler J, Windle K, Borremans M, Resseler S, Van Roey J, Parys W, Vangeneugden T, Van Baelen B, Rosenberg Z; Ring Study Team. Safety and Efficacy of a Dapivirine Vaginal Ring for HIV Prevention in Women. N Engl J Med. 2016 Dec 1;375(22):2133-2143. doi: 10.1056/NEJMoa1602046. PMID 27959766

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened between 27 March 2012 and 22 Oct 2014. The IPM 027 trial was originally designed with a sample size of approximately 1,650 participants, which was increased to approximately 1,950 participants according to the amended protocol (Protocol Version 1.0 Amendment 3.0, dated 12 September 2013).
  Participants were recruited and enrolled at 6 RCs in South Africa and 1 RC in Uganda. A total of 3,425 participants were screened, of whom 1,959 participants were enrolled.
Pre-assignment Details: Participants who provided written informed consent at Screening Visit 1 were invited to undergo screening assessments for the trial. Participant screening was conducted over two scheduled Screening Visits with a maximum window period of 28 days between the two visits.
Period: Overall Study
Arm/Group | Placebo Vaginal Ring | Dapivirine Vaginal Ring
Started | 652 | 1307
Completed (A number of completed participants rolled over to the open-label extension of this trial (IPM 032, NCT02862171)) | 435 (107 participants rolled over to the open-label extension of the trial) | 902 (238 participants rolled over to the open-label extension of the trial)
Not Completed | 217 | 405
Not completed — Withdrawal by Subject | 24 | 54
Not completed — Lost to Follow-up | 20 | 54
Not completed — Death | 1 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Pregnancy | 13 | 29
Not completed — inappropriate enrollment | 0 | 1
Not completed — Multiple Reasons | 3 | 1
Not completed — not HIV seroconversion-related | 93 | 176
Not completed — HIV seroconversion-related | 55 | 80
Not completed — Non-compliance | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Vaginal Ring | Dapivirine Vaginal Ring | Total
Number analyzed (Participants) | 652 | 1307 | 1959
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (5.92) | 25.9 (5.85) | 26.0 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 652 | 1307 | 1959
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 642 | 1299 | 1941
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  South Africa | 587 | 1175 | 1762
  Uganda | 65 | 132 | 197
BMI [Mean (Standard Deviation); unit: kg/(m^2)] | 28.2 (6.80) | 28.1 (7.12) | 28.1 (7.01)
Education level [Count of Participants; unit: Participants]
  secondary education | 371 | 775 | 1146
  primary education | 228 | 384 | 612
  tertiary education | 29 | 90 | 119
  unknown | 24 | 58 | 82
Marital status [Count of Participants; unit: Participants]
  Never married | 581 | 1166 | 1747
  Married | 63 | 118 | 181
  Legally separated | 7 | 13 | 20
  Widowed | 0 | 8 | 8
  Divorced | 1 | 2 | 3
Has children [Count of Participants; unit: Participants] | 601 | 1190 | 1791
Has main sex partner [Count of Participants; unit: Participants] | 640 | 1284 | 1924
Usual number of vaginal sex act each month [Mean (Standard Deviation); unit: vaginal sex acts per month] — Population: Only this number of participants provided a response.
  vaginal sex acts per month
    number analyzed (Participants) | 625 | 1248 | 1873
    (all) | 8.4 (10.46) | 8.1 (10.32) | 8.2 (10.37)

OUTCOME MEASURES:

1. Primary Outcome: HIV-1 Seroconversion According to Comprehensive HIV Testing Algorithm.
Description: HIV-1 seroconversion measured by rapid and specialised laboratory testing according to the comprehensive HIV testing algorithm.
Time Frame: 24 months
Population: This population consisted of all participants included in the ITT population (all randomised), excluding those who were not identified as HIV-seropositive at the Enrollment Visit, but who were later found to be already HIV-1 infected at enrollment through HIV-1 RNA PCR testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo Vaginal Ring
Number analyzed (Participants) | 1302 | 650
Participants | 82 | 61

2. Primary Outcome: All Adverse Events
Description: Self-reports, physical examination, gynaecological assessments, including pelvic/speculum examination, laboratory tests and other indicated investigations. All AEs will be reported, regardless of grade or relatedness.
Time Frame: 24 months
Population: The safety population included all participants who had been randomized to IP and used at least one DVR or placebo ring.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo Vaginal Ring
Number analyzed (Participants) | 1306 | 652
Participants | 1147 | 561

3. Secondary Outcome: The Incidence Rate of HIV-2 Seroconversion.
Description: Rapid and specialised laboratory testing according to the comprehensive HIV testing algorithm in Appendix C of protocol.
Time Frame: 24 months
Population: This population consisted of all participants included in the ITT population, excluding those who were not identified as HIV-seropositive at the Enrollment Visit, but who were later found to be already HIV-1 infected at enrollment through HIV-1 RNA PCR testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo Vaginal Ring
Number analyzed (Participants) | 1302 | 650
Participants | 0 | 0

4. Secondary Outcome: The Incidence of Curable STIs
Description: The percentage of participants testing positive for any STI (gonorrhoea, chlamydia, trichomonas, syphilis) will be assessed.
Time Frame: 24 months
Population: The safety population included all participants who had been randomized to IP and used at least one DVR or placebo ring.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo Vaginal Ring
Number analyzed (Participants) | 1271 | 624
Participants | 682 | 315

5. Secondary Outcome: Percentage of Participants With Pregnancy in Each Trial Arm Over the IP Use Period;
Description: The percentage of participants with pregnancies in each treatment group. For each treatment group, the numerator will include the number of participants that had a positive urine pregnancy test during the trial period.
Time Frame: 24 months
Population: The safety population included all participants who had been randomized to IP and used at least one DVR or placebo ring.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo Vaginal Ring
Number analyzed (Participants) | 1306 | 652
Participants | 43 | 20

6. Secondary Outcome: The Percentage of Women Who Report Adherence to the Use of the Vaginal Ring Inserted Once Every 4 Weeks Over the Trial Period;
Description: Questionnaires and qualitative data regarding sexual behaviour and adherence to the use of a vaginal ring inserted once every 4 weeks over the trial period.
  Dapivirine residual levels in used rings and dapivirine plasma concentrations are two objective measures of adherence to DVR ring use,
Time Frame: 24 months
Population: The objective measures (dapivirine residual levels in used rings and dapivirine plasma concentrations) used can only be determined for participants who used the active vaginal dapivirine ring.
Measure: Number; unit: percentage of participants with data
Arm/Group | Dapivirine Vaginal Ring
Number analyzed (Participants) | 1302
percentage of participants with data
  Week 4: number analyzed (Participants) | 1276
  Week 4 | 77.1
  Week 8: number analyzed (Participants) | 1254
  Week 8 | 76.5
  Week 12: number analyzed (Participants) | 1236
  Week 12 | 75.0
  Week 16: number analyzed (Participants) | 1208
  Week 16 | 74.9
  Week 20: number analyzed (Participants) | 1192
  Week 20 | 73.7
  Week 24: number analyzed (Participants) | 1176
  Week 24 | 73.9
  Week 28: number analyzed (Participants) | 1162
  Week 28 | 73.4
  Week 32: number analyzed (Participants) | 1151
  Week 32 | 73.5
  Week 36: number analyzed (Participants) | 1141
  Week 36 | 74.9
  Week 40: number analyzed (Participants) | 1133
  Week 40 | 76.1
  Week 44: number analyzed (Participants) | 1116
  Week 44 | 76.3
  Week 48: number analyzed (Participants) | 1093
  Week 48 | 77.4
  Week 52: number analyzed (Participants) | 1073
  Week 52 | 78.5
  Week 56: number analyzed (Participants) | 1051
  Week 56 | 78.9
  Week 60: number analyzed (Participants) | 1025
  Week 60 | 81.1
  Week 64: number analyzed (Participants) | 1008
  Week 64 | 82.7
  Week 68: number analyzed (Participants) | 982
  Week 68 | 85.0
  Week 72: number analyzed (Participants) | 957
  Week 72 | 83.9
  Week 76: number analyzed (Participants) | 917
  Week 76 | 84.0
  Week 80: number analyzed (Participants) | 871
  Week 80 | 81.4
  Week 84: number analyzed (Participants) | 831
  Week 84 | 81.1
  Week 88: number analyzed (Participants) | 790
  Week 88 | 81.5
  Week 92: number analyzed (Participants) | 743
  Week 92 | 81.6
  Week 96: number analyzed (Participants) | 708
  Week 96 | 83.1
  Week 100: number analyzed (Participants) | 682
  Week 100 | 82.6
  Week 104: number analyzed (Participants) | 680
  Week 104 | 80.1

7. Secondary Outcome: The Percentage of Women Who Report the Use of the Vaginal Ring as Acceptable;
Description: Questionnaires and qualitative data regarding the acceptability of use of a vaginal ring inserted once every 4 weeks over the trial period; Number of participants with positive response. Response of 'likely' or 'very likely' to the question: 'If in the future a vaginal ring was available that provided some protection against HIV, and it was similar to the one you used in this trial, how likely would you be to keep it inserted in your vagina every day?'
Time Frame: 24 months
Population: as for outcome 3
Measure: Number; unit: percentage of participants with data
Arm/Group | Dapivirine Vaginal Ring | Placebo Vaginal Ring
Number analyzed (Participants) | 1302 | 650
percentage of participants with data
  Week 4 | 97.4 | 98.7
  Week 24 | 98.7 | 98.6

8. Secondary Outcome: The Percentage of Participants With HIV-1 Drug Resistance Mutations Among Participants Who Acquire HIV-1.
Description: The analysis of HIV-1 drug resistance will be primarily descriptive in nature, and will depend on the pattern of resistance mutations observed in the HIV-1 seroconverters. The proportion of HIV-1 seroconverters with at least one HIV-1 drug resistant mutation will be presented overall, and by treatment arm, with corresponding 95% CIs.
Time Frame: 24 months
Population: The virology population included all ITT participants with seroconversion, excluding those who never received investigational product, or were retrospectively found to be HIV-1 RNA positive at enrollment (m-ITT) or were HIV-1 infected after discontinuation of ring use. Seroconversions among participants who were continued on open-label DVR-004 were included in the DVR-004 group, independent of initial randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo Vaginal Ring
Number analyzed (Participants) | 87 | 61
Participants | 84 | 58

ADVERSE EVENTS:
Time Frame: 4 years and 9 months During the double-blind treatment period, the median (range) number of days of ring exposure was 764.0 (28 - 826) days in participants in the DVR group and 763.5 (8 - 839) days in participants in the placebo ring group.
Arm/Group | Placebo Vaginal Ring | Dapivirine Vaginal Ring
All-Cause Mortality (participants affected / at risk) | 3/652 | 2/1306
Serious Adverse Events (participants affected / at risk) | 9/652 | 41/1306
Other Adverse Events (participants affected / at risk) | 561/652 | 1147/1306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Vaginal Ring (N=652) | Dapivirine Vaginal Ring (N=1306)
Febrile Infection (Infections and infestations) | 0 (0) | 3 (3)
Malaria (Infections and infestations) | 0 (0) | 3 (3)
Acute Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Injection site abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acral lentiginous melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Vaginal Ring (N=652) | Dapivirine Vaginal Ring (N=1306)
Gynaecological chlamydia infection (Infections and infestations) | 213 (328) | 427 (669)
Genital infection female (Infections and infestations) | 126 (166) | 300 (388)
Genitourinary tract gonococcal infection (Infections and infestations) | 108 (146) | 252 (333)
Upper respiratory tract infection (Infections and infestations) | 115 (247) | 231 (536)
Trichomoniasis (Infections and infestations) | 103 (150) | 225 (351)
Urinary tract infection (Infections and infestations) | 100 (151) | 185 (261)
Vulvovaginal candidiasis (Infections and infestations) | 84 (110) | 174 (258)
Vulvovaginitis (Infections and infestations) | 72 (132) | 115 (251)
Vaginitis bacterial (Infections and infestations) | 39 (50) | 99 (129)
Viral rhinitis (Infections and infestations) | 35 (64) | 73 (148)
Nasopharyngitis (Infections and infestations) | 29 (30) | 66 (73)
Malaria (Infections and infestations) | 30 (43) | 61 (93)
Viral upper respiratory tract infection (Infections and infestations) | 24 (32) | 47 (58)
Gastroenteritis (Infections and infestations) | 19 (22) | 47 (53)
Cervicitis (Infections and infestations) | 21 (26) | 29 (31)
Vulvovaginitis trichomonal (Infections and infestations) | 17 (24) | 33 (44)
Pelvic inflammatory disease (Infections and infestations) | 26 (28) | 21 (25)
Pharyngitis (Infections and infestations) | 16 (19) | 31 (34)
Metrorrhagia (Reproductive system and breast disorders) | 193 (335) | 353 (616)
Menorrhagia (Reproductive system and breast disorders) | 71 (112) | 135 (231)
Dysmenorrhoea (Reproductive system and breast disorders) | 51 (95) | 90 (127)
Cervical dysplasia (Reproductive system and breast disorders) | 47 (56) | 88 (98)
Menometrorrhagia (Reproductive system and breast disorders) | 42 (60) | 87 (122)
Pelvic pain (Reproductive system and breast disorders) | 25 (26) | 71 (78)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 21 (23) | 45 (49)
Vulval ulceration (Reproductive system and breast disorders) | 24 (29) | 33 (47)
Diarrhoea (Gastrointestinal disorders) | 44 (64) | 64 (76)
Gastritis (Gastrointestinal disorders) | 29 (57) | 53 (102)
Abdominal Pain Lower (Gastrointestinal disorders) | 19 (19) | 41 (46)
Constipation (Gastrointestinal disorders) | 22 (24) | 38 (42)
Abdominal Pain (Gastrointestinal disorders) | 16 (17) | 30 (32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (58) | 79 (126)
Myalgia (Musculoskeletal and connective tissue disorders) | 39 (69) | 74 (107)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (31) | 53 (57)
Headache (Nervous system disorders) | 77 (95) | 112 (139)
Soft tissue injury (Injury, poisoning and procedural complications) | 17 (17) | 26 (26)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 30 (35)

LIMITATIONS AND CAVEATS:
Dapivirine residual levels in used rings and dapivirine plasma concentrations are two objective measures of adherence to DVR ring use; however, they were found to be an imperfect measure of adherence as they cannot distinguish different patterns of use during the month. In addition, self-reported adherence based on the adherence questionnaires was also considered to have limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No